CLINICAL TRIAL: NCT00382018
Title: A Randomized Phase III Trial to Test the Strategy of Changing Therapy Versus Maintaining Therapy for Metastatic Breast Cancer Patients Who Have Elevated Circulating Tumor Cell Levels at First Follow-Up Assessment
Brief Title: S0500 Treatment Decision Making Based on Blood Levels of Tumor Cells for Metastatic Breast Cancer Treated With Chemo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000504319; S0500 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Active Comparator): Patients continue to receive regular treatment without change at the discretion of the physician. Patients are eligible for other first-line chemotherapy trials. No further blood is collected.
  Interventions: Drug: chemotherapy
- Group 2 (Experimental): Patients continue to receive their current chemotherapy regimen without change.
  Interventions: Drug: chemotherapy
- Group 3, Arm I (Active Comparator): Patients continue with their current chemotherapy regimen without change.
  Interventions: Drug: chemotherapy
- Group 3, Arm II (Experimental): Patients switch to a different chemotherapy regimen. Selection of a new chemotherapy regimen is made by the patient's doctor.
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: chemotherapy — No administration details available

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Measuring blood levels of tumor cells may help in learning how well chemotherapy works to kill metastatic breast cancer cells and allow doctors to plan better treatment. When blood levels of tumor cells are high while receiving chemotherapy, it is not yet known whether it is more effective to change chemotherapy regimens at that time or wait until disease progression.

PURPOSE: This randomized phase III trial is studying treatment decision making based on blood levels of tumor cells in women with metastatic breast cancer receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether women with metastatic breast cancer and elevated circulating tumor cells (CTCs) (≥ 5 per 7.5 mL of whole blood) after 3 weeks of first-line chemotherapy derive increased overall survival from changing to an alternative chemotherapy regimen at the next course rather than waiting for clinical evidence of progressive disease before changing to an alternative chemotherapy regimen.
* Determine whether these patients derive increased progression-free survival (PFS) from changing to an alternative chemotherapy regimen at the next course rather than waiting for clinical evidence of progressive disease before changing to an alternative chemotherapy regimen.
* Confirm previous findings that patients with < 5 CTCs per 7.5 mL of whole blood on initial screening have longer median OS and PFS than patients with ≥ 5 CTCs per 7.5 mL of whole blood.
* Determine the prognostic value of sequentially collected CTC values in these patients.
* Compare toxicity between patients with and without elevated CTCs after 3 weeks of first-line chemotherapy AND between the two randomized treatment arms.

Secondary

* Compare the prognostic and predictive value of CTC number vs breast cancer tumor markers, including CA 15-3 and carcinoembryonic antigen.
* Create a serum specimen bank for future biologic investigation.

OUTLINE: This is a partially blinded, partially randomized, multicenter study. Patients are assigned to 1 of 3 groups based on circulating tumor cells (CTCs) after 1 course of chemotherapy.

All patients undergo blood collection before their first dose of first-line chemotherapy* to determine baseline CTC count. Patients with < 5 CTCs at baseline are assigned to group I. Patients with ≥ 5 CTCs at baseline undergo a second blood draw on day 22 (after completion of 1 course of chemotherapy). Patients with < 5 CTCs after completing 1 course of chemotherapy are assigned to group 2. Patients with ≥ 5 CTCs after completion of 1 course of chemotherapy are assigned to group 3.

NOTE: *Chemotherapy may be initiated while waiting for the baseline CTC result.

* Group 1 (low risk of early progression): Patients continue to receive regular treatment without change at the discretion of the physician. Patients are eligible for other first-line chemotherapy trials. No further blood is collected.
* Group 2 (moderate risk of early progression): Patients continue to receive their current chemotherapy regimen without change.
* Group 3 (high risk of early progression): Patients are stratified according to HER-2 status (positive vs negative) and disease type (bone-only vs measurable disease). Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients continue with their current chemotherapy regimen without change.
  * Arm II: Patients switch to a different chemotherapy regimen. Selection of a new chemotherapy regimen is made by the patient's doctor.

Patients receiving hormonal therapy or biologic therapy and chemotherapy continue to receive the hormonal or biologic therapy unchanged regardless of CTC level.

In groups 2 and 3, blood is collected periodically during chemotherapy and then at the completion of chemotherapy. Samples are examined for CTCs via the CellSearch™ blood test. Blood is also tested for CA 15-3 and carcinoembryonic antigen (CEA).

After completion of study therapy, patients are followed for up to 5 years.

PROJECTED ACCRUAL: A total of 500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Clinical evidence of metastatic disease (stage IV disease)
  * Newly metastatic disease OR progressive metastatic disease while on hormonal therapy
* Meets 1 of the following criteria:

  * Measurable disease
  * Bone-only disease* NOTE: *Patients with nonmeasurable disease that does not include bone are not eligible
* HER-2 status determined by immunohistochemistry (IHC) or fluorescent in situ hybridization (FISH) assay

  * HER-2 positivity is defined as IHC 3+ or FISH+
  * If IHC is indeterminate (2+), FISH must be performed to classify disease
* Planning to undergo first-line chemotherapy for metastatic disease
* Patients with brain metastases must have stable disease for > 90 days after completion of prior radiotherapy to the brain
* No leptomeningeal disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Zubrod performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or stage I or II cancer currently in complete remission

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior hormonal therapy, bisphosphonate therapy, trastuzumab (Herceptin®), and/or bevacizumab for metastatic disease allowed

  * Any number of exogenous hormonal therapies for metastatic disease and/or as adjuvant therapy allowed
* At least 1 year since prior adjuvant chemotherapy
* At least 2 weeks since prior minor surgery and recovered
* At least 4 weeks since prior major surgery and recovered
* No prior chemotherapy for metastatic disease
* Concurrent hormonal therapy and/or bisphosphonate therapy allowed
* Concurrent trastuzumab and/or bevacizumab allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2006-10; Primary Completion 2015-12 (Actual); Study Completion 2017-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B. Smerage, MD, PhD, Study Chair — University of Michigan Rogel Cancer Center; Daniel F. Hayes, MD, Study Chair — University of Michigan Rogel Cancer Center; Eric P. Winer, MD, Study Chair — Dana-Farber Cancer Institute
Locations (296):
- United States (296):
  - Regional Medical Center, Anniston, Alabama
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Providence Cancer Center, Anchorage, Alaska
  - NEA Medical Center - Stadium Boulevard, Jonesboro, Arkansas
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - California Cancer Care, Incorporated - Greenbrae, Greenbrae, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Stanford Cancer Center, Stanford, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Regional Cancer Care at Community Hospital North, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Mercy Hospital, Portland, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Saint Vincent Hospital at Worcester Medical Center, Worcester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Clemens Regional Medical Center, Mount Clemens, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center at Carrie J. Babb Cancer Center, Bolivar, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - UMDNJ University Hospital, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - Presbyterian Cancer Treatment Center at Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center - South, Las Cruces, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Dickstein Cancer Treatment Center at White Plains Hospital Center, White Plains, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Granville Medical Center, Oxford, North Carolina
  - Duke Health Raleigh Hospital, Raleigh, North Carolina
  - Person Memorial Hospital, Roxboro, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Cleveland Clinic Beachwood Family Health and Surgery Center, Beachwood, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Cleveland Clinic Foundation - Strongsville, Strongsville, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - St. Charles Medical Center - Bend, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Providence Cancer Center at PMCC, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Ephrata Cancer Center at Ephrata Community Hospital, Ephrata, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Cancer Center at Phoenixville Hospital, Phoenixville, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Cancer Centers of the Carolinas - Easley, Easley, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Virginia Cancer Institute - West End, Richmond, Virginia
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Oncology Alliance, SC - Milwaukee - West, Wauwatosa, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Derived] Smerage JB, Barlow WE, Hortobagyi GN, Winer EP, Leyland-Jones B, Srkalovic G, Tejwani S, Schott AF, O'Rourke MA, Lew DL, Doyle GV, Gralow JR, Livingston RB, Hayes DF. Circulating tumor cells and response to chemotherapy in metastatic breast cancer: SWOG S0500. J Clin Oncol. 2014 Nov 1;32(31):3483-9. doi: 10.1200/JCO.2014.56.2561. Epub 2014 Jun 2. PMID 24888818

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 624 patients were registered for screening. 29 patients were excluded due to initial CTC test not completed(17) and ineligible(12). 276 did not have increased CTC levels (Arm A). 319 patients had increased CTC levels. Additional 31 patients were excluded from 319 due to no CTC values on Day 21. Thus total 288 patients in ArmB, ArmC2 and ArmC2.
Groups:
- Arm A (Baseline CTCs < 5, Low Risk): Patients did not have increased CTCs at baseline (defined as five or more CTCs per 7.5 mL WB). Patients would be treated at clinician's discretion. Patients could be enrolled in other trials while being followed. Patients were followed only for overall survival (OS) and progression-free survival (PFS).
- Arm B (Baseline CTCs >= 5, Day 22 CTCs < 5, Moderate Risk): Patients had increased CTCs at baseline (defined as five or more CTCs per 7.5 mL WB) but < 5 CTCs at first follow-up (Day 22). Patients would maintain current therapy and will not be randomized.
- Arm C1 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk): Patients had increased CTCs at baseline (defined as five or more CTCs per 7.5 mL WB) and >= 5 CTCs at first follow-up (Day 22). Patients would be randomized to maintain current therapy.
- Arm C2 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk): Patients had increased CTCs at baseline (defined as five or more CTCs per 7.5mL WB) and >= 5CTCs at first follow-up (Day22). Patients would be randomized to change therapy to a different drug or combination of drugs.
Period: Overall Study
Arm/Group | Arm A (Baseline CTCs < 5, Low Risk) | Arm B (Baseline CTCs >= 5, Day 22 CTCs < 5, Moderate Risk) | Arm C1 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk) | Arm C2 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk)
Started (Patients in this group were only followed for OS and PFS. Thus, no treatment status data.) | 276 | 165 | 64 | 59
Completed | 276 (This group of patients did not receive protocol treatment.) | 0 | 0 | 0
Not Completed | 0 | 165 | 64 | 59
Not completed — Progression | 0 | 136 | 51 | 43
Not completed — Death | 0 | 9 | 7 | 11
Not completed — Withdrawal by Subject | 0 | 4 | 3 | 4
Not completed — Other, not protocol specified | 0 | 16 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Baseline CTCs < 5, Low Risk) | Arm B (Baseline CTCs >= 5, Day 22 CTCs < 5, Moderate Risk) | Arm C1 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk) | Arm C2 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk) | Total
Number analyzed (Participants) | 276 | 165 | 64 | 59 | 564
Age, Customized [Count of Participants; unit: Participants]
  Age 55 years or older | 163 | 94 | 38 | 39 | 334
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 276 | 165 | 64 | 59 | 564
  Male | 0 | 0 | 0 | 0 | 0
Black Race [Count of Participants; unit: Participants] | 50 | 23 | 15 | 7 | 95
Measurable disease [Count of Participants; unit: Participants] — Measurable disease: Lesions that can be accurately measured in at least one dimension by 1) medical photograph (skin or oral lesion), palpation, plain x-ray, CT, MRI or other conventional technique with longest diameter 2 cm or greater in the axial plane (bone lesions not included), or 2) spiral CT with longest diameter 1 cm or greater. Ultrasound is suitable only for superficial disease (superficial palpable nodes, subcutaneous lesions, thyroid nodules).
  Participants | 221 | 137 | 47 | 50 | 455
No. of patients classified by disease subtype [Count of Participants; unit: Participants] | 275 | 162 | 64 | 59 | 560
Homo receptor positive, HER2 negative [Count of Participants; unit: Participants] — Population: Only patients classified by disease subtype category will be included in the analysis.
  Participants
    number analyzed (Participants) | 275 | 162 | 64 | 59 | 560
    (all) | 148 | 93 | 50 | 39 | 330
Triple negative [Count of Participants; unit: Participants] — Population: Only patients classified by disease subtype category will be included in the analysis.
  Participants
    number analyzed (Participants) | 275 | 162 | 64 | 59 | 560
    (all) | 74 | 33 | 11 | 16 | 134
HER2 positive [Count of Participants; unit: Participants] — Population: Only patients classified by disease subtype category will be included in the analysis.
  Participants
    number analyzed (Participants) | 275 | 162 | 64 | 59 | 560
    (all) | 53 | 36 | 3 | 4 | 96

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Every 3 months until progression then every 6 months for 5 years or until death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm C1 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk) | Arm C2 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk)
Number analyzed (Participants) | 64 | 59
months | 10.7 [9.1 to 14.8] | 12.5 [8.4 to 16.3]
Statistical Analysis 1: Comparison: Arm C1 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk) vs Arm C2 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk); Hazard Ration of overall survival compared Arm C2 to Arm C1; Test type: Superiority or Other; p = 0.98, Log Rank; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.69 to 1.47]

2. Primary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: every 3 months until progression. From date of registration to date of first documentation of progressive disease, death due to any cause or symptomatic deterioration, whichever occurs first, assessed up to five years.
Population: Three patients in Arm C2 were judged as progression on day 22 and were excluded from the PFS analysis but were included in the OS analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm C1 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk) | Arm C2 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk)
Number analyzed (Participants) | 64 | 56
months | 3.5 [2.1 to 4.7] | 4.6 [3.1 to 6.7]
Statistical Analysis 1: Comparison: Arm C1 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk) vs Arm C2 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk); Hazard Ratio of progression free survival compared Arm C2 to Arm C1; Test type: Superiority or Other; p = 0.64, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.64 to 1.32]

3. Primary Outcome: Overall Survival
Description: as for outcome 1
Time Frame: Every 3 months until progression then every 6 months for 5 years or until death
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm C (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk): Patients had increased CTCs at baseline (defined as five or more CTCs per 7.5 mL WB) and >= 5 CTCs at first follow-up (Day 22). Patients would be randomized to maintain current therapy or change therapy to an alternative therapy
Arm/Group | Arm A (Baseline CTCs < 5, Low Risk) | Arm B (Baseline CTCs >= 5, Day 22 CTCs < 5, Moderate Risk) | Arm C (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk)
Number analyzed (Participants) | 276 | 165 | 123
months | 35 [29 to 38.5] | 23 [19 to 28.3] | 13 [10.2 to 15.0]

4. Primary Outcome: Progression Free Survival
Description: From date of registration to date of first documentation of progressive disease, death due to any cause or symptomatic deterioration, whichever occurs first. Patients last known to be alive and progression-free are censored at date of last contact.
Time Frame: every 3 months until progression
Population: Three patients in Arm C were judged as progressing on day 22 and were excluded from the PFS analysis but were included in the OS analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Baseline CTCs < 5, Low Risk) | Arm B (Baseline CTCs >= 5, Day 22 CTCs < 5, Moderate Risk) | Arm C (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk)
Number analyzed (Participants) | 276 | 165 | 120
months | 11.1 [9.5 to 12.5] | 8.9 [8.1 to 10.8] | 4.9 [3.8 to 5.7]

5. Secondary Outcome: Number of Patients With Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 3.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Toxicity assessment was evaluated after 3 weeks, 6 weeks, and every 6 weeks thereafter until progression
Population: Patients in 'Arm A (Baseline CTCs < 5, Low Risk)' were followed only for overall survival (OS) and progression-free survival (PFS). Adverse events were not collected/assessed in these patients. And only patients who were evaluable for Adverse Event Assessment were included in the following analysis results.
Measure: Number; unit: Participants
Arm/Group | Arm B (Baseline CTCs >= 5, Day 22 CTCs < 5, Moderate Risk) | Arm C1 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk) | Arm C2 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk)
Number analyzed (Participants) | 161 | 64 | 56
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 8 | 1 | 3
  AST, SGOT | 10 | 1 | 6
  Albumin, serum-low (hypoalbuminemia) | 5 | 2 | 4
  Alkaline phosphatase | 7 | 5 | 8
  Allergic reaction/hypersensitivity | 3 | 1 | 1
  Allergic rhinitis | 2 | 1 | 1
  Allergy/Immunology-Other (Specify) | 1 | 0 | 1
  Anorexia | 16 | 5 | 9
  Ascites (non-malignant) | 0 | 1 | 1
  Auditory/Ear-Other (Specify) | 0 | 1 | 0
  Bilirubin (hyperbilirubinemia) | 5 | 2 | 3
  Blood/Bone Marrow-Other (Specify) | 1 | 1 | 0
  CNS cerebrovascular ischemia | 1 | 0 | 0
  Calcium, serum-high (hypercalcemia) | 2 | 1 | 0
  Calcium, serum-low (hypocalcemia) | 5 | 3 | 4
  Confusion | 2 | 0 | 1
  Constipation | 12 | 5 | 6
  Constitutional Symptoms-Other (Specify) | 1 | 0 | 0
  Cough | 3 | 0 | 0
  Creatinine | 15 | 5 | 2
  Dehydration | 17 | 6 | 7
  Dermatology/Skin-Other (Specify) | 2 | 1 | 2
  Diarrhea | 55 | 10 | 15
  Distention/bloating, abdominal | 0 | 1 | 0
  Dizziness | 2 | 2 | 1
  Dry eye syndrome | 0 | 0 | 1
  Dry mouth/salivary gland (xerostomia) | 1 | 0 | 1
  Dry skin | 5 | 1 | 1
  Dyspnea (shortness of breath) | 18 | 9 | 9
  Edema: head and neck | 2 | 0 | 0
  Edema: limb | 3 | 0 | 6
  Fatigue (asthenia, lethargy, malaise) | 103 | 36 | 36
  Febrile neutropenia | 6 | 0 | 2
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 3 | 3 | 1
  Flatulence | 1 | 0 | 0
  Flushing | 2 | 0 | 0
  Gastrointestinal-Other (Specify) | 1 | 0 | 0
  Glucose, serum-high (hyperglycemia) | 13 | 4 | 7
  Glucose, serum-low (hypoglycemia) | 0 | 0 | 1
  Hair loss/Alopecia (scalp or body) | 20 | 5 | 5
  Heartburn/dyspepsia | 2 | 1 | 0
  Hemoglobin | 100 | 32 | 38
  Hemorrhage, Respiratory tract NOS | 1 | 0 | 0
  Hemorrhage, GI - Stomach | 1 | 0 | 0
  Hemorrhage, GU - Uterus | 1 | 0 | 0
  Hemorrhage, pulmonary/upper respiratory - Nose | 7 | 4 | 0
  Hot flashes/flushes | 3 | 1 | 4
  Hyperpigmentation | 1 | 3 | 0
  Hypertension | 6 | 0 | 2
  Hypotension | 3 | 1 | 1
  Ileus, GI (functional obstruction of bowel) | 0 | 1 | 0
  Induration/fibrosis (skin and subcutaneous tissue) | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 1 | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 0 | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - UTI | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Nose | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Oral cav | 0 | 1 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Sinus | 3 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Skin | 0 | 0 | 2
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 3 | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Up airway | 1 | 0 | 0
  Infection with unknown ANC - Sinus | 1 | 0 | 0
  Infection with unknown ANC - Skin (cellulitis) | 2 | 0 | 0
  Infection with unknown ANC - Urinary tract NOS | 0 | 2 | 0
  Infection-Other (Specify) | 2 | 0 | 0
  Injection site reaction/extravasation changes | 0 | 0 | 1
  Insomnia | 2 | 1 | 1
  Left ventricular systolic dysfunction | 1 | 0 | 1
  Leukocytes (total WBC) | 28 | 11 | 10
  Lymphopenia | 8 | 2 | 3
  Magnesium, serum-low (hypomagnesemia) | 2 | 0 | 1
  Memory impairment | 0 | 1 | 0
  Metabolic/Laboratory-Other (Specify) | 1 | 1 | 0
  Mood alteration - anxiety | 2 | 0 | 1
  Mood alteration - depression | 3 | 1 | 1
  Mucositis/stomatitis (clinical exam) - Oral cavity | 10 | 0 | 2
  Mucositis/stomatitis (functional/symp) - Oral cav | 2 | 2 | 1
  Muscle weakness, not d/t neuropathy - Extrem-lower | 2 | 0 | 0
  Muscle weakness, not d/t neuropathy - Extrem-upper | 1 | 0 | 0
  Muscle weakness, not d/t neuropathy - body/general | 1 | 1 | 5
  Musculoskeletal/Soft Tissue-Other (Specify) | 1 | 1 | 0
  Nail changes | 2 | 1 | 3
  Nasal cavity/paranasal sinus reactions | 1 | 0 | 0
  Nausea | 27 | 10 | 10
  Neuropathy: motor | 1 | 0 | 0
  Neuropathy: sensory | 23 | 3 | 5
  Neutrophils/granulocytes (ANC/AGC) | 71 | 23 | 25
  Ocular/Visual-Other (Specify) | 0 | 0 | 1
  Osteonecrosis (avascular necrosis) | 0 | 0 | 1
  Pain - Abdomen NOS | 0 | 2 | 1
  Pain - Back | 6 | 1 | 3
  Pain - Bladder | 1 | 0 | 0
  Pain - Bone | 27 | 8 | 9
  Pain - Breast | 0 | 1 | 0
  Pain - Chest wall | 1 | 0 | 0
  Pain - Chest/thorax NOS | 3 | 0 | 1
  Pain - Extremity-limb | 0 | 0 | 2
  Pain - Face | 1 | 0 | 0
  Pain - Head/headache | 5 | 2 | 1
  Pain - Joint | 8 | 1 | 4
  Pain - Muscle | 10 | 0 | 2
  Pain - Neck | 0 | 0 | 1
  Pain - Neuralgia/peripheral nerve | 1 | 0 | 0
  Pain - Oral cavity | 1 | 0 | 0
  Pain - Oral-gums | 0 | 0 | 1
  Pain - Pain NOS | 2 | 0 | 1
  Pain - Pelvis | 1 | 0 | 0
  Pain - Rectum | 1 | 0 | 0
  Pain - Scalp | 0 | 1 | 0
  Pain - Stomach | 0 | 1 | 1
  Pain - Throat/pharynx/larynx | 1 | 0 | 0
  Pain - Vagina | 1 | 0 | 0
  Pain-Other (Specify) | 0 | 3 | 1
  Phosphate, serum-low (hypophosphatemia) | 1 | 1 | 2
  Platelets | 42 | 16 | 23
  Pleural effusion (non-malignant) | 0 | 0 | 1
  Pneumonitis/pulmonary infiltrates | 2 | 0 | 0
  Potassium, serum-high (hyperkalemia) | 1 | 0 | 0
  Potassium, serum-low (hypokalemia) | 4 | 1 | 1
  Proteinuria | 2 | 0 | 0
  Pruritus/itching | 2 | 0 | 0
  Pulmonary/Upper Respiratory-Other (Specify) | 1 | 0 | 0
  Rash/desquamation | 2 | 0 | 2
  Rash: acne/acneiform | 2 | 2 | 0
  Rash: hand-foot skin reaction | 10 | 4 | 3
  Renal/Genitourinary-Other (Specify) | 1 | 0 | 0
  Restrictive cardiomyopathy | 2 | 0 | 0
  Retinopathy | 0 | 0 | 1
  Rigors/chills | 1 | 1 | 0
  SVT and nodal arrhythmia - Atrial tachycardia/PAT | 1 | 0 | 0
  SVT and nodal arrhythmia - Sinus tachycardia | 3 | 0 | 0
  Sodium, serum-high (hypernatremia) | 1 | 0 | 1
  Sodium, serum-low (hyponatremia) | 6 | 0 | 2
  Sweating (diaphoresis) | 1 | 0 | 1
  Syndromes-Other (Specify) | 0 | 0 | 1
  Taste alteration (dysgeusia) | 6 | 2 | 2
  Thrombosis/thrombus/embolism | 5 | 1 | 2
  Thyroid function, high | 0 | 1 | 0
  Triglyceride, serum-high (hypertriglyceridemia) | 0 | 1 | 0
  Urinary frequency/urgency | 1 | 0 | 0
  Vaginal dryness | 0 | 1 | 0
  Vision-blurred vision | 1 | 1 | 0
  Vomiting | 38 | 10 | 14
  Watery eye (epiphora, tearing) | 1 | 1 | 0
  Weight loss | 8 | 2 | 3

6. Other Pre Specified Outcome: Correlation of CTC Levels With Breast Cancer Tumor Markers
Time Frame: Baseline, Weeks 4, 8, 13, 25, 37 and at progression
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Toxicity assessment was evaluated after 3 weeks, 6 weeks, and every 6 weeks thereafter until progression
Description: Patients in 'Arm A (Baseline CTCs < 5, Low Risk)' were followed only for overall survival (OS) and progression-free survival (PFS). Adverse events were not collected/assessed in these patients. Only patients who were evaluable for Adverse Event Assessment were included in the analysis result.
Arm/Group | Arm B (Baseline CTCs >= 5, Day 22 CTCs < 5, Moderate Risk) | Arm C1 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk) | Arm C2 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk)
Serious Adverse Events (participants affected / at risk) | 0/161 | 1/64 | 0/56
Other Adverse Events (participants affected / at risk) | 152/161 | 57/64 | 53/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm B (Baseline CTCs >= 5, Day 22 CTCs < 5, Moderate Risk) (N=161) | Arm C1 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk) (N=64) | Arm C2 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk) (N=56)
Gastrointestinal-Other (Gastrointestinal disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Renal/Genitourinary-Other (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm B (Baseline CTCs >= 5, Day 22 CTCs < 5, Moderate Risk) (N=161) | Arm C1 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk) (N=64) | Arm C2 (Baseline CTCs >= 5, Day 22 CTCs >= 5, High Risk) (N=56)
Hemoglobin (Blood and lymphatic system disorders) | 112 | 35 | 43
Constipation (Gastrointestinal disorders) | 20 | 8 | 8
Diarrhea (Gastrointestinal disorders) | 66 | 15 | 16
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 11 | 0 | 2
Nausea (Gastrointestinal disorders) | 30 | 10 | 11
Pain - Abdomen NOS (Gastrointestinal disorders) | 4 | 5 | 2
Vomiting (Gastrointestinal disorders) | 52 | 17 | 17
Edema: limb (General disorders) | 15 | 2 | 8
Fatigue (asthenia, lethargy, malaise) (General disorders) | 112 | 40 | 42
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 7 | 4 | 2
Pain - Pain NOS (General disorders) | 3 | 1 | 3
Pain-Other (General disorders) | 5 | 4 | 4
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 2 | 1 | 3
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 13 | 5 | 3
AST, SGOT (Investigations) | 17 | 5 | 10
Alkaline phosphatase (Investigations) | 14 | 7 | 10
Bilirubin (hyperbilirubinemia) (Investigations) | 11 | 3 | 7
Creatinine (Investigations) | 24 | 8 | 7
Leukocytes (total WBC) (Investigations) | 29 | 11 | 10
Lymphopenia (Investigations) | 9 | 2 | 3
Metabolic/Laboratory-Other (Investigations) | 3 | 1 | 3
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 77 | 24 | 28
Platelets (Investigations) | 49 | 19 | 25
Weight loss (Investigations) | 10 | 4 | 3
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 8 | 3 | 6
Anorexia (Metabolism and nutrition disorders) | 19 | 5 | 11
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 4 | 1 | 3
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 9 | 4 | 7
Dehydration (Metabolism and nutrition disorders) | 27 | 8 | 10
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 22 | 7 | 7
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6 | 4 | 4
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 8 | 1 | 4
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 2 | 1 | 6
Pain - Back (Musculoskeletal and connective tissue disorders) | 20 | 4 | 6
Pain - Bone (Musculoskeletal and connective tissue disorders) | 64 | 21 | 20
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 7 | 1 | 3
Pain - Joint (Musculoskeletal and connective tissue disorders) | 18 | 4 | 7
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 14 | 3 | 3
Dizziness (Nervous system disorders) | 6 | 2 | 3
Neuropathy: sensory (Nervous system disorders) | 28 | 4 | 7
Pain - Head/headache (Nervous system disorders) | 8 | 5 | 5
Mood alteration - anxiety (Psychiatric disorders) | 4 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 5 | 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 53 | 18 | 20
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 20 | 5 | 6
Nail changes (Skin and subcutaneous tissue disorders) | 2 | 1 | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 | 0 | 3
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 10 | 4 | 3
Hot flashes/flushes (Vascular disorders) | 4 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less